CLINICAL TRIAL: NCT01501682
Title: Long Term Complaints After Elective Repair for Small Umbilical or Epigastric Hernias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Liv Erritzøe-Jervild, stud.med, Zealand University Hospital
Other Study IDs: ventralexmesh_KoegeHospital
Record Dates: First submitted 2011-12-18; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Ventral Hernia
Keywords: ventralex; ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- primary suture: operated with primary suture
- other mesh: operated with insertion of another mesh
- ventralex: operated with insertion of ventralex mesh

SUMMARY:
The purpose of this study is to compare the long-term complaints after ventral hernia repair after insertion of different types of mesh compared with primary suture. Also recurrence of hernia will be discussed.

DETAILED DESCRIPTION:
The purpose of this study is to compare the long-term complaints after ventral hernia repair after insertion of different types of mesh compared with primary suture. Based on a questionnaire selected patients will be invited to clinical examination for recurrence and more detailed interview.

ELIGIBILITY:
Inclusion Criteria:

* operated for ventral hernia from the year 2004 to the year 2009

Exclusion Criteria:

* liver cirrhosis
* pregnancy
* combined hernia
* operation for ventral hernia and other operation
* laparoscopic operation
* acute operation
* recurrence of hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: operated for ventral hernia from the year 2004 to the year 2009 at Koege Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liv Erritzøe-Jervild, Principal Investigator — Køge Hospital
Locations (2):
- Denmark (2):
  - Koege hospital, Koege
  - Køge sygehus, Køge

REFERENCES:
- [Derived] Erritzoe-Jervild L, Christoffersen MW, Helgstrand F, Bisgaard T. Long-term complaints after elective repair for small umbilical or epigastric hernias. Hernia. 2013 Apr;17(2):211-5. doi: 10.1007/s10029-012-0960-z. Epub 2012 Jul 14. PMID 22797701